CLINICAL TRIAL: NCT02595476
Title: The Influence of Depth of Anesthesia on Pupillary Reactivity to a Standardized Stimulus Under Steady-state Remifentanil Analgesia
Brief Title: Influence of Depth of Anesthesia on Pupillary Reactivity to a Standardized Stimulus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, Pr Isabelle CONSTANT, Professor Isabelle COnstant, Hôpital Armand Trousseau
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Anesthésie Trousseau 002
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Pain
Keywords: analgesia; pupillometry; general anesthesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Remifentanil; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS 55 (Experimental): 1. Induction:
     TCI propofol (6 µg/ml) - remifentanil (4 ng/ml) Atracurium IV (0.5 mg/kg)
  2. Orotracheal Intubation
  3. Remifentanil target decreased to 1 ng/ml
  4. Propofol target adjustment to reach BIS 55
  5. 10 minutes steady state
  6. Tetanic stimulation (ulnar nerve): 100 Hz, 60 milliamps, 5 seconds
  7. Pupillary dilation recording (videopupillometer Algiscan)
  Interventions: Drug: Remifentanil; Drug: propofol; Device: TCI; Procedure: Tetanic stimulation; Device: Algiscan
- BIS 25 (Active Comparator): 1. Induction:
     TCI propofol (6 µg/ml) - remifentanil (4 ng/ml) Atracurium IV (0.5 mg/kg)
  2. Orotracheal Intubation
  3. Remifentanil target decreased to 1 ng/ml
  4. Propofol target adjustment to reach BIS 25
  5. 10 minutes steady state
  6. Tetanic stimulation (ulnar nerve): 100 Hz, 60 milliamps, 5 seconds
  7. Pupillary dilation recording (videopupillometer Algiscan)
  Interventions: Drug: Remifentanil; Drug: propofol; Device: TCI; Procedure: Tetanic stimulation; Device: Algiscan

INTERVENTIONS:
Drug: Remifentanil
Drug: propofol
Device: TCI
Procedure: Tetanic stimulation
Device: Algiscan — Pupillometry

SUMMARY:
A standardized tetanic stimulation is applied to patients under propofol-remifentanil TCI, in a cross-over fashion, at two different levels of anesthesia monitored by the BIS: BIS 25 and BIS 55. Remifentanil target remains constant during the whole study period (1 ng/ml). Pupillary reflex dilation is recorded after each stimulation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* scheduled for an idiopathic scoliosis surgical correction

Exclusion Criteria:

* Ophtalmologic pathology
* Neurologic or muscular pathology
* Metabolic pathology
* Chronic pain

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Post-stimulation Pupillary reflex dilation | 30 seconds
  percentage of dilation compared to pre-stimulation pupillary diameter

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, MD, PHD, Study Director — Hopital Armand Trousseau
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France

REFERENCES:
- [Derived] Sabourdin N, Peretout JB, Khalil E, Guye ML, Louvet N, Constant I. Influence of Depth of Hypnosis on Pupillary Reactivity to a Standardized Tetanic Stimulus in Patients Under Propofol-Remifentanil Target-Controlled Infusion: A Crossover Randomized Pilot Study. Anesth Analg. 2018 Jan;126(1):70-77. doi: 10.1213/ANE.0000000000001802. PMID 28107273